CLINICAL TRIAL: NCT02852291
Title: Parents Make the Difference II: A Randomized Experiment of a Parent Training Program for Caregivers of Young Children Designed to Reduce the Use of Harsh Punishment and Improve Child-caregiver Relationships
Brief Title: Parents Make the Difference II: Trial of a Parenting Intervention
Acronym: PMD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: International Rescue Committee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-1111
Record Dates: First submitted 2016-03-07; First posted 2016-08-02 (Estimated); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Parenting; Child Abuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Parents Make the Difference (Experimental): Parents Make the Difference (Caregivers attend 10 group parent training sessions)
  Interventions: Behavioral: Parents Make the Difference
- Parents Make the Difference Plus (Experimental): Parents Make the Difference Plus (Caregivers attend 10 group parent training sessions and receive 3 home visits)
  Interventions: Behavioral: Parents Make the Difference Plus
- Waitlist Control (No Intervention): No parenting intervention until the end of the study period

INTERVENTIONS:
Behavioral: Parents Make the Difference — 10 parent training sessions delivered to groups of caregivers
  Arms: Parents Make the Difference
Behavioral: Parents Make the Difference Plus — 10 parent training sessions delivered to groups of caregivers, with 3 home visits
  Arms: Parents Make the Difference Plus

SUMMARY:
Multisite randomized trial of a parenting intervention in Liberia for caregivers of young children. Two main objectives of the "Parents Make the Difference" program are to teach parents (a) skills for decreasing harsh punishments and replacing those with positive ways to manage children's behavior and (b) skills for having more positive interactions with their children, including interactions that encourage learning. As a result of positive changes in parenting, the investigators expect that, over time, children's behavioral and cognitive well-being will improve and that future abuse and poor developmental outcomes will be prevented in the long-term.

DETAILED DESCRIPTION:
This is a multisite randomized trial of a parenting intervention in Liberia for caregivers of young children. The "Parents Make the Difference" program is designed to teach parents (a) skills for decreasing harsh punishments and replacing those with positive ways to manage children's behavior and (b) skills for having more positive interactions with their children. As a result of positive changes in parenting, the investigators expect that, over time, children's behavioral and cognitive well-being will improve and that the intervention will prevent future abuse and poor developmental outcomes in the long-term. This study will randomize 816 caregivers of children ages 3 or 4 years to 1 of 3 study arms: standard group program, group program plus home visits, waitlist control.

ELIGIBILITY:
Inclusion Criteria:

* caregiver of child ages 3 or 4
* live within catchment area of each study site
* caregiver is at least 18 years old

Exclusion Criteria:

* does not live with child

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Caregiver use of harsh discipline practices; assessed using Discipline Interview, Locally-derived items | 1 month post treatment
  Extent to which caregivers engage in harsh discipline practices
Parent-Child Interactions (Parental Acceptance-Rejection Questionnaire; Locally-derived items assessing positive interactions) | 1 month post treatment
  Quality of parent-child relationships and interactions

SECONDARY OUTCOMES:
Caregiver use of harsh discipline practices; assessed using Discipline Interview, Locally-derived items | 12 months post treatment
  Use of harsh discipline practices, including physical and verbal strategies
Parent-Child Interactions (Parental Acceptance-Rejection Questionnaire; Locally-derived items assessing positive interactions) | 12 months post treatment
  Quality of parent-child relationships and interactions
Child social-emotional development and functioning: Ages and Stages Questionnaire; Strengths and Difficulties Questionnaire: emotion problems and peer problems subscales | 1 and 12 months post treatment
  Indicators of child emotional problems and problems in peer relationships
Child behavior: Locally-derived measure of disruptive/non-compliant behaviors; Strengths and Difficulties Questionnaire (conduct problems subscale) | 1 and 12 months post treatment
  Frequency of disruptive behaviors / SDQ items related to behavioral problems
Parental Stress: Parental Stress Scale | 1 and 12 months post treatment
  Level of caregiver parenting-related stress
Parental knowledge of child development: Locally-derived scale | 1 and 12 months post treatment
  Locally relevant indicators of parental knowledge about child development
Marital relationship quality: selected items from Conflict Tactics Scale and locally-derived scale of marital relationship quality | 1 and 12 months post treatment
  Indicators of quality of marital interactions, including relationship violence
Caregiver mental health: General Health Questionnaire (subscale A), Patient Health Questionnaire-9 | 1 and 12 months post treatment
  Indicators of caregiver mental health symptoms
Handwashing Behavior Indicators (e.g., access to hand washing station) | 1 and 12 months post treatment
  Basic indicators of hand washing behavior and resources
Child cognitive skills (verbal ability); assessed with a story comprehension task and instruction-following task | 1 and 12 months post treatment
  Child verbal abilities (brief assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Puffer, PhD, Principal Investigator — Duke University
Locations (1):
- International Rescue Committee, Monrovia, Liberia

IPD SHARING:
Plan to Share IPD: Yes
following anonymization and publication